CLINICAL TRIAL: NCT01331317
Title: The Effect of Paricalcitol Versus Placebo on Plasma N-Terminal-proBNP in Patients With Type 1 Diabetes Mellitus and Diabetic Nephropathy
Brief Title: Effect of a Vitamin D Analogue vs Placebo on p-NT-proBNP in Patients With Type 1 DM and Diabetic Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peter Rossing (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Peter Rossing, Senior Physician, DMSc, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-011255-44
Record Dates: First submitted 2010-07-27; First posted 2011-04-08 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Disease; Diabetic Nephropathy
Keywords: Cardiovascular disease and mortality; Plasma NTproBNP; UAER
MeSH Terms: conditions — Cardiovascular Diseases; Diabetic Nephropathies | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paricalcitol (Other): Crossover study between paricalcitol and placebo
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Paricalcitol — capsule, 1-2 micrograms daily for 90 days
  Other Names: Zemplar

SUMMARY:
The primary objective is to assess the impact of three months of treatment with an active vitamin D analogue on a risk marker for excess overall mortality and cardiovascular morbidity/mortality in Type 1 diabetic patients with diabetic kidney disease. The hypothesis is that active vitamin D analogue treatment reduces the risk of cardiovascular morbidity and mortality in patients with type 1 diabetic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Type 1 diabetes mellitus
* Diabetic nephropathy (defined by persistent albuminuria, > 300 mg/24 hr or 200µg/min in 2 of 3 consecutive samples, presence of diabetic retinopathy and absence of clinical or laboratory evidence of other kidney or renal tract disease
* Chronic kidney disease stage 3 and 4
* S-Parathyroid hormone (s-PTH)> 35pg/ml
* Stabile RAAS-blocking and diuretic treatment

Exclusion Criteria:

* Other kidney disease than diabetic nephropathy
* Myocardial infarction within the last three months prior to visit 1
* Coronary artery revascularization within the last three months prior to visit 1
* Transitional cerebral ischemia (TCI) or apoplexia within the last three months prior to visit 1
* Cardiac Failure (NYHA Class III or IV)
* Kidney Failure (GFR <15ml/min), dialysis, kidney transplantation)
* Liver disease with serum alanine aminotransferase (ALT>3 x the normal value
* Alcohol/drug abuse
* Hypercalcemia (serum ionized calcium >1.35 mmol /L)
* Medication with phosphate and/or vitamin D-containing medications, which can not be paused during the study
* Clinical signs of vitamin D toxicity
* Pregnant or nursing women
* Fertile women not using chemical or mechanical (IUD) contraceptive methods
* Current disulfiram treatment
* Allergy to the study drug
* Patient unable to understand the informed consent
* Any other condition or therapy which, in the opinion of the investigator, makes the patient not suited for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in plasma NT-proBNP | 7 months

SECONDARY OUTCOMES:
Change in Glomerular Filtration Rate (GFR) | 7 months
Change in Urinary Albumin Excretion Rate | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Lise Tarnow, MD, Principal Investigator — Steno Diabetes Center A/S
Locations (1):
- Steno Diabetes Center A/S, Gentofte Municipality, Denmark